CLINICAL TRIAL: NCT06620510
Title: A Multicenter, Retrospective Data Analysis Study on the Long-term Survival Rate of the 'Immuncell-LC Goups' and 'Non-treatment Groups' in Patient Undergo Curative Resection (PEIT, RFA or Operation) for Hepatocellular Carcinoma in Korea
Brief Title: Retrospective Study of Long-Term Survival of "Immuncell-LC" in Patients Undergoing Curative Resection for HCC in Korea
Status: Completed | Type: Observational
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IIC-I03
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- No intervention: Patients who were in non-treatment group in phase 3 clinical trial IIC-I01(NCT00699816).
  Interventions: Biological: No Interventions
- Immuncell-LC Group: Patients who were in Immuncell-LC group in phase 3 clinical trial IIC-I01(NCT00699816).
  Interventions: Biological: Immuncell-LC

INTERVENTIONS:
Biological: Immuncell-LC — Activated T lymphocyte
  Groups: Immuncell-LC Group
Biological: No Interventions — Patients who were in non-treatment group in phase 3 clinical trial IIC-I01(NCT00699816).
  Groups: No intervention

SUMMARY:
To observation that long term follow-up study of 'Immuncell-LC groups' and 'Non-treatment groups' in patient undergo curative resection (PEIT, RFA or Operation) for hepatocellular carcinoma in Korea

DETAILED DESCRIPTION:
The purpose of this study is to retrospectively compare the long-term survival of patients who participated in the "Randomized, open-label, multicenter phase 3 clinical trial to evaluate the efficacy and safety of Immunocel-LC treatment and no treatment in Korean patients with hepatocellular carcinoma (HCC) who received potentially curative treatment [surgical resection, radiofrequency ablation (RFA), or percutaneous ethanol injection (PEI)] (NCT00699816). HCC was diagnosed by pathological evaluation or radiological imaging studies. Eligibility criteria also included hepatic function of Child-Pugh class A and an Eastern Cooperative Oncology Group performance status score of 0 or 1. Exclusion criteria included autoimmune disease or immunodeficiency, previous or current malignant tumor other than HCC, and severe allergic disorders. Pregnant or breastfeeding women and women planning to become pregnant were also excluded. All eligible participants were randomly assigned to receive adjuvant immunotherapy using a CIK cell agent (the immunotherapy group) or no adjuvant treatment (control group) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients of participated in the(ClinicalTrials.gov Identifier:NCT00699816)clinical trial.

Exclusion Criteria:

* NA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This long term follow-UP study is observation about the Immuncell-LC Groups' and 'Non-treatment Groups' in patient undergo curative resection (PEIT, RFA or Operation) for Hepatocelluar Carcinoma in Korea.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Recurrence-free Survival(RFS) | up to 9 years
  RFS was measured from the date of randomization to the first recurrence or to death from any cause.
  Radiological test should be operated by dynamic CT, dynamic MRI or by angiography.

SECONDARY OUTCOMES:
Overall Survival(OS) | up to 9 years
  Overall survival was measured from the date of randomization until death from any cause. And OS was estimated using Kaplan-Meier methods with 95% confidence intervals (CIs).
Cancer-specific Survivals(CSS) | up to 9 years
  Cancer-specific survival was measured from the date of randomization until death resulting from HCC.

CONTACTS AND LOCATIONS:
Overall Officials: JinHee Kang, Study Director — Global Product Development Division
Locations (1):
- Seoul National University Hospital, Seoul, South Korea